CLINICAL TRIAL: NCT00356746
Title: A Prospective, Randomized Trial to Study the Effects of Different Anesthetic Agents on the Perioperative Immune Response
Brief Title: Inflammatory Response During Anesthesia and Surgery
Acronym: IRAS
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: European Association of Cardiothoracic Anaesthesiologists (Unknown)
Responsible Party: WF Buhre, UMC Utrecht, Department of Anesthesiology
Other Study IDs: METC-05/261-E
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Systemic Inflammatory Response Syndrome; Myocardial Ischemia
Keywords: Perioperative inflammatory response; General anesthesia; Toll-Like Receptors
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Full blood smaples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: elective CABG only patients
- 2: elective ICD replacement surgical patients requiring general anesthesia

SUMMARY:
The purpose of this study is to investigate the effects of total intravenous anesthesia versus volatile anesthesia on the perioperative inflammatory response during and after major surgery.

DETAILED DESCRIPTION:
Patients undergoing major surgical procedures, in particular those undergoing cardiac surgery, develop a severe inflammatory response in up to 50% of cases leading to increased mortality and morbidity. The inflammatory response depends on the surgical procedure and on patient related factors like genetic predisposition and co morbidities. However, in vitro studies showed that the type and duration of general anaesthesia also influences the extent of perioperative inflammation.

Comparison: total intravenous anesthesia by propofol is compared to volatile anesthesia by isoflurane with respect to development of perioperative inflammatory response.

The IRAS study is a single centre study, executed in the University Medical Centre Utrecht, The Netherlands. Four different patient groups are included. 1) Patients undergoing coronary artery bypass grafting (CABG) with use of cardiopulmonary bypass (CPB), 2) patients undergoing aorta aneurysm repair via endovascular approach and 3) via conventional open procedure, and 4) patients undergoing surgery for replacement of implantable cardioverter defibrillator (ICD).

The IRAS is a prospective, randomized clinical trial. Patients are randomly assigned to a intravenous or a balanced anaesthesia technique. Peripheral blood samples are drawn before, during and up to 72h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and planned for elective Coronary Artery Bypass Grafting (CABG), aorta surgery or Implantable Cardioverter Defibrillator (ICD) replacement

Exclusion Criteria:

* Emergency operations
* Patients undergoing combined or re-do procedures
* Patients who are diagnosed with or undergoing treatment for a steroid or hormone disorder, excluding diabetes
* Patients suffering from chronic inflammatory diseases
* Patients suffering form current infections
* Patients currently treated with steroids
* Patients undergoing treatment or care for a malignancy
* Patients participating in another study that may interfere with the endpoints of the IRAS trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: specific surgical patients receiving general anesthesia of university teaching hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Perioperative inflammatory response through measurement of expression and responsiveness of Toll-like Receptor (TLR) 2 and 4 of monocytes from full blood samples. | 72 hours

SECONDARY OUTCOMES:
Parameters of systemic haemodynamics | 72 hours
Need of vasoactive medication to develop predefined haemodynamic goals | 72 hours
Biochemical parameter of myocardial ischaemia and infarction (Troponin-I), measured immediately before and after surgery, 24 hr and 72hr after surgery | 72 hours
Serious adverse events assessed 3 days after surgery, at discharge, 30 days and one year after surgery | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cor J Kalkman, Prof MD PhD, Study Chair — University Medical Centre Utrecht, The Netherlands; Wolfgang F Buhre, MD PhD, Study Director — University Medical Centre Utrecht, The Netherlands; Gerard Pasterkamp, Prof MD PhD, Study Director — University Medical Centre Utrecht, The Netherlands
Locations (1):
- UMC Utrecht, Division of Perioperative Care and Emergency Medicine, Department of Anesthesiology, Utrecht, Netherlands

REFERENCES:
- [Background] de Kleijn D, Pasterkamp G. Toll-like receptors in cardiovascular diseases. Cardiovasc Res. 2003 Oct 15;60(1):58-67. doi: 10.1016/s0008-6363(03)00348-1. PMID 14522407
- [Background] de Rossi LW, Brueckmann M, Rex S, Barderschneider M, Buhre W, Rossaint R. Xenon and isoflurane differentially modulate lipopolysaccharide-induced activation of the nuclear transcription factor KB and production of tumor necrosis factor-alpha and interleukin-6 in monocytes. Anesth Analg. 2004 Apr;98(4):1007-1012. doi: 10.1213/01.ANE.0000106860.27791.44. PMID 15041589
- [Background] Larsen B, Hoff G, Wilhelm W, Buchinger H, Wanner GA, Bauer M. Effect of intravenous anesthetics on spontaneous and endotoxin-stimulated cytokine response in cultured human whole blood. Anesthesiology. 1998 Nov;89(5):1218-27. doi: 10.1097/00000542-199811000-00023. PMID 9822011
- [Derived] Flier S, Concepcion AN, Versteeg D, Kappen TH, Hoefer IE, de Lange DW, Pasterkamp G, Buhre WF. Monocyte hyporesponsiveness and Toll-like receptor expression profiles in coronary artery bypass grafting and its clinical implications for postoperative inflammatory response and pneumonia: An observational cohort study. Eur J Anaesthesiol. 2015 Mar;32(3):177-88. doi: 10.1097/EJA.0000000000000184. PMID 25405275
- [Derived] Flier S, Post J, Concepcion AN, Kappen TH, Kalkman CJ, Buhre WF. Influence of propofol-opioid vs isoflurane-opioid anaesthesia on postoperative troponin release in patients undergoing coronary artery bypass grafting. Br J Anaesth. 2010 Aug;105(2):122-30. doi: 10.1093/bja/aeq111. Epub 2010 Jun 23. PMID 20573633